CLINICAL TRIAL: NCT03410459
Title: Long-term Adverse Effects After Laparoscopic Sleeve Gastrectomy and Roux en Y Gastric Bypass (Part A)
Brief Title: Long-term Adverse Effects After Bariatric Surgery on Bone Density
Acronym: FUB-A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: FUB Study Bone
Record Dates: First submitted 2018-01-02; First posted 2018-01-25 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Morbid Obesity
MeSH Terms: conditions — Obesity, Morbid | interventions — Absorptiometry, Photon

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gastric Bypass (Active Comparator): Patients ≥ 5 years after laparoscopic gastric bypass receive DEXA (= Dual-energy x-ray absorptiometry) in order to measure bone mass density
  Interventions: Diagnostic Test: DEXA (= Dual-energy x-ray absorptiometry)
- Sleeve gastrectomy (Active Comparator): Patients ≥ 5 years after laparoscopic sleeve gastrectomy receive DEXA (= Dual-energy x-ray absorptiometry) in order to measure bone mass density
  Interventions: Diagnostic Test: DEXA (= Dual-energy x-ray absorptiometry)

INTERVENTIONS:
Diagnostic Test: DEXA (= Dual-energy x-ray absorptiometry) — measurement of vertebral bone and hip bone mineral density

SUMMARY:
The goal of this trial is to examine long-term effects of laparoscopic gastric bypass (LRYGB) and sleeve gastrectomy (LSG) on bone mineral density, fracture risk, and body composition ≥ 5 years post-surgery.

DETAILED DESCRIPTION:
Bariatric surgery shows impressive results in terms of weight loss and resolution of comorbidities. Still, there are questions as to the frequency of long-term adverse effects: data on alterations in bone health are missing,

The goal of this trial is to examine long-term effects of laparoscopic gastric bypass (LRYGB) and sleeve gastrectomy (LSG) on bone mineral density, fracture risk, and body composition ≥ 5 years post-surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received laparoscopic sleeve gastrectomy (LSG) or laparoscopic gastric bypass (LRYGB) ≥ 5 years ago as a primary bariatric procedure will be eligible for this study.

Exclusion Criteria:

* LSG or LRYGB as a secondary bariatric procedure (e.g. after gastric banding), patients receiving secondary bariatric operation after LSG resp LRYGB (e.g. biliopancreatic diversion), pregnancy (due to radiation exposition)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2018-02-02 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
Total hip T-Score measured with dual-energy x-ray absorptiometry | 5-7 years after bariatric surgery
  measured score will be compared to reference score for this age

SECONDARY OUTCOMES:
Total vertebral T-Score measured with dual-energy x-ray absorptiometry | 5-7 years after bariatric surgery
  measured score will be compared to reference score for this age
fracture risk assessed by FRAX score | 5-7 years after bariatric surgery
  measured score will be compared to reference score for this age
plasma concentration of C-terminal telopeptide (CTX) | 5-7 years after bariatric surgery
  measured plasma concentration will be compared to reference for this age
plasma concentration of vitamin D3 | 5-7 years after bariatric surgery
  measured plasma concentration will be compared to reference for this age

CONTACTS AND LOCATIONS:
Overall Officials: Bettina K Wölnerhanssen, MD, Principal Investigator — Clinical Research St. Claraspital Basel
Locations (1):
- St Claraspital, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No